CLINICAL TRIAL: NCT03018834
Title: Anakinra Versus Placebo Double Blind Randomized Controlled Trial for the Treatment of Acute MyocarditIS
Brief Title: Anakinra Versus Placebo for the Treatment of Acute MyocarditIS
Acronym: ARAMIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P150921; 2016-003433-20 (EudraCT Number)
Record Dates: First submitted 2016-12-12; First posted 2017-01-12 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Acute Myocarditis
Keywords: Acute Myocarditis; ANAKINRA
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: ANAKINRA (Experimental): ANAKINRA 100 mg/daily subcutaneously once a day until hospital discharge, for a maximum of 14 days, in addition to standard care: ACE and Beta-blocker for 6 months.
  Interventions: Drug: ANAKINRA 100 mg/daily subcutaneously
- B: Placebo (Placebo Comparator): PLACEBO 100 mg/daily subcutaneously once a day until hospital discharge, for a maximum of 14 days, in addition to standard care: ACE and Beta-blocker for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANAKINRA 100 mg/daily subcutaneously — ANAKINRA 100 mg/daily subcutaneously once a day until hospital discharge, for a maximum of 14 days, in addition to standard care: ACE and Beta-blocker for 6 months.
  Other Names: Kineret
  Arms: A: ANAKINRA
Drug: Placebo — PLACEBO 100 mg/daily subcutaneously once a day until hospital discharge, for a maximum of 14 days, in addition to standard care: ACE and Beta-blocker for 6 months.
  Arms: B: Placebo

SUMMARY:
There is no specific treatment of acute myocarditis, especially during the inflammatory period. Interleukin (IL) is specifically involved during this period and play a role in myocardial oedema. ANAKINRA, an IL-1β Blocker, is a new treatment that has never been evaluated in myocarditis. The benefit for the patient could be important with a reduction of heart failure and ventricular arrhythmias.

Hypothesis : ANAKINRA in addition to standard therapy for treatment of Acute Myocarditis is superior to standard therapy based on an association of beta-blockers and Angiotensin-Converting-Enzyme inhibitor (ACE).

DETAILED DESCRIPTION:
It is a Double Blind Randomized clinical trial Phase IIb of superiority, enrolling two groups: one group treated with the standard of care, defined as the maximum tolerated dosage of any beta blockers and ACE, and placebo versus ANAKINRA in addition to the standard of care in patients treated for an acute Myocarditis.

Patients will be randomized to receive ANAKINRA 100 mg/daily or placebo subcutaneously once a day until hospital discharge, for a maximum of 14 days, in addition to standard care: ACE and Beta-blocker for 6 months. Randomization 1:1 will be conducted centrally using the electronic Case Report Form (eCRF).

As an exploratory analysis, a second randomization for ACE discontinuation in patients without left ventricular dysfunction (LVEF > 50%) at one month post discharge will be performed.

One group will stopped the treatment at one month and the second group will continued the ACE for 6 months. This second randomization is in open label.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for Acute myocarditis defined as:
* Chest Pain (or modification of the ECG) AND Troponin Rise (*1.5 Normal range) AND Myocarditis proven by MRI in the first 72h after admission
* Age > 18 and <65 years old
* Accepting effective contraception during treatment duration (men and women childbearing potential)
* Signed informed consent Normal Coronary angiography or coronary CT Scan (made during the previous year is acceptable) (normal is defined as stenosis < 50%) (In the case of patients under 40 with typical MRI of myocarditis, coronary angiography is not mandatory and left to the doctor's discretion)

Exclusion Criteria:

* Active coronary disease
* Clinical Suspicion or proven underlying disease: systemic lupus, antiphospholipid antibodies, Lyme disease, trypanosomiase disease, myositis, signs of sarcoidosis, giant cell myocarditis, treated chronic inflammatory disease, tuberculosis, HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV), Hepatitis B virus (HBV) infection,
* Latex allergy
* Pregnancy, breastfeeding
* Contra-indication to ANAKINRA (known hypersensitivity to the active substance or to any of the excipients, neutropenia < 1,5.10^9/L)
* Renal failure, Creatine Clearance (CrCl) < 30 ml/min (MDRD)
* Malignancy or any comorbidity limiting survival or conditions predicting inability to complete the study
* History of malignancy
* Non Steroidian Anti Inflammatory drug within the past 14 days
* Anti Tumor Necrosis Factor (TNF) within the past 14 days
* No affiliation to the French Health Care System "sécurité sociale"
* Hepatic impairment = Child-Pugh Class C
* Mechanical ventilation
* Circulatory assistance

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of days alive free of any myocarditis complications | within 28 days post hospitalization
  Number of days alive free of any myocarditis complications defined as ventricular arrhythmias, heart failure, chest pain, ventricular dysfunction defined as LVEF<50%, within 28 days post hospitalization

SECONDARY OUTCOMES:
Total cost | on average 14 days
  Total cost
Total Quality Adjusted Life Year (QALYs), | on average 14 days
  measure of the perceived utility by patients of a medication (Anakinra) that corresponds to a year of life gained
Incremental cost effectiveness | on average 14 days
  cost-effectiveness of ANAKINRA in the setting of acute myocarditis
Cost utility ratios | on average 14 days
  Cost utility ratios
Left Ventricul Ejection Fraction (LVEF) assessed by cardiac Magnetic Resonance Imaging (MRI) | at 6 month
  Left Ventricul Ejection Fraction (LVEF) assessed by cardiac Magnetic Resonance Imaging (MRI)
Left Ventricul Ejection Fraction (LVEF) assessed by Trans Thoracic Echocardiograhy (TTE) | at 6 month
  Left Ventricul Ejection Fraction (LVEF) assessed by Trans Thoracic Echocardiograhy (TTE)
LVEF assessed by cardiac MRI | at 1 year
  LVEF assessed by cardiac MRI
LVEF assessed by cardiac TTE | at 1 year
  LVEF assessed by cardiac TTE
All cause of death rate | during the 12 months follow-up
  All cause of death rate
Cardiovascular death | at 12 months
  Cardiovascular death
Heart Failure | at 12 months
  Heart Failure
Ventricular tachycardia | during the 12 months follow-up
  Ventricular tachycardia
NT-proBNP above 450 pg/mL (in patients aged below 50); above 900 pg/mL (age 50-75 years) or BNP ≤ 400pg/mL 50% decrease of the troponin level at discharge compared to admission | at Day0
  NT-proBNP above 450 pg/mL (in patients aged below 50); above 900 pg/mL (age 50-75 years) or BNP ≤ 400pg/mL 50% decrease of the troponin level at discharge compared to admission
NT-proBNP above 450 pg/mL (in patients aged below 50); above 900 pg/mL (age 50-75 years) or BNP ≤ 400pg/mL 50% decrease of the troponin level at discharge compared to admission | an average of 14 days
  NT-proBNP above 450 pg/mL (in patients aged below 50); above 900 pg/mL (age 50-75 years) or BNP ≤ 400pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu KERNEIS, MD, Principal Investigator — ACTION Study Group - Assistance Publique - Hôpitaux de Paris; Fleur COHEN AUBART, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Gilles MONTALESCOT, MD, PhD, Study Director — ACTION Study Group - Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - ACTION Study Group - Department of Cardiology - Pitié Salpétrière Hospital, 47 Bd de l'Hopital, Paris
  - Department of internal medicine - Pitié Salpétrière Hospital, 47 Bd de l'Hopital, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Werner B, Roznowska-Wojtowicz A, Puchalski M. Diagnosis and Management of Pediatric Myocarditis. Pediatr Infect Dis J. 2025 Mar 1;44(3):e95-e98. doi: 10.1097/INF.0000000000004678. Epub 2024 Dec 17. No abstract available. PMID 39705605
- [Derived] Kerneis M, Cohen F, Combes A, Amoura Z, Pare C, Brugier D, Puymirat E, Abtan J, Lattuca B, Dillinger JG, Hauguel-Moreau M, Silvain J, Salem JE, Gandjbakhch E, Hekimian G, Redheuil A, Vicaut E, Montalescot G; ACTION Study Group. Rationale and design of the ARAMIS trial: Anakinra versus placebo, a double blind randomized controlled trial for the treatment of acute myocarditis. Arch Cardiovasc Dis. 2023 Oct;116(10):460-466. doi: 10.1016/j.acvd.2023.07.004. Epub 2023 Aug 12. PMID 37640625